CLINICAL TRIAL: NCT06245148
Title: The Effect of Intraoperative Ephedrine Use on the Incidence of Hypothermia After Major Surgery
Status: Completed | Type: Observational
Sponsor: Acibadem University (Other)
Responsible Party: Principal Investigator, Lerzan Doğan, Dr, Acibadem University
Other Study IDs: 2023-14/506
Record Dates: First submitted 2024-01-15; First posted 2024-02-07 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Ephedrine Usage and Hypothermia Incidence; Effects of Ephedrine on Thermogulation
Keywords: Ephedrine usage; Intraoperative hypotension; Intraoperative hypothermia;; Major surgery
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hypothermia
  Interventions: Other: Observation
- Normothermia
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — Observation

SUMMARY:
Intraoperative hypothermia is a common and potentially severe complication during major surgical procedures. The consequences of intraoperative hypothermia can be far-reaching, affecting patient outcomes, recovery times, and overall healthcare costs. Therefore, strategies aimed at preventing hypothermia are of paramount importance in modern surgical practice. However, despite all the measures taken, some patients may still become hypothermic at the end of surgery. Understanding these factors can enhance the quality of daily practice. Medications used intraoperatively can decrease the threshold for vasoconstriction, and some of them have been reported to influence thermoregulation. For example, ephedrine is a sympathomimetic amine used to maintain hemodynamic stability, but there is a report about its thermogenic effect. One study found that patients who received an intraoperative infusion of ephedrine had a significantly lower decrease in core temperature and these patients had a more stable hemodynamic profile. It was employed in obese patients for its thermogenic and appetite-suppressing effects until its adverse effects prevented its use. Ephedrine has an unintended yet significant effect on body temperature regulation, which has raised questions about its role in contributing to the incidence of hypothermia in the postoperative period. The purpose of this study is to investigate the potential relationship between the intraoperative use of ephedrine and the incidence of hypothermia following major surgery.

DETAILED DESCRIPTION:
This study aims to investigate the potential relationship between the intraoperative use of ephedrine and the incidence of hypothermia following major surgery. The primary goal is to determine the effect of intraoperative ephedrine use on the incidence of hypothermia after major surgery. The secondary goal is to identify patient characteristics associated with an increased risk of hypothermia despite all measures taken. The results of this study could have important implications for the quality of care for patients undergoing major surgery.

ELIGIBILITY:
Inclusion Criteria:

* all adult patients (age 18 years) who received ephedrine during general anesthesia undergoing major surgical procedures

Exclusion Criteria:

* Patients undergoing minor surgical procedures
* Patients scheduled for day surgeries
* Patients patients (those under the age of 18)
* Patients with a history of thyroid disease
* Patients undergoing brain surgery
* Patients undergoing radiological interventions,
* Trauma patients
* Patients directly transferred from the intensive care unit to the operating room
* Patients with preoperative fever (either low or high)
* Patients who have received vasoactive agents within 24 hours before surgery
* Patients with sepsis and/or septic shock, or fever within a week before surgery
* Patients who have received vasoactive agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This observational study was conducted over a span of four years, from January 2020 to 2023,
Sampling Method: Probability Sample
Enrollment: 9259 (Actual)
Dates: Start 2019-01-02 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Incidence of Hypothermia after Major Surgery | From anesthesia induction until discharge to a ward, with the event defined as the time the patient meets all discharge criteria, assessed up to 10 hours post-operatively.
  The occurrence of hypothermia in patients who have undergone major surgery, specifically comparing those who received intraoperative ephedrine to those who did not.

SECONDARY OUTCOMES:
Patient Characteristics Associated with Increased Hypothermia Risk | From anesthesia induction until discharge to a ward, with the event defined as the time the patient meets all discharge criteria, assessed up to 10 hours post-operatively.
  Specific patient characteristics or factors that may increase the risk of hypothermia despite the implementation of measures to prevent it

CONTACTS AND LOCATIONS:
Locations (1):
- Acibadem University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Matsukawa T, Sessler DI, Sessler AM, Schroeder M, Ozaki M, Kurz A, Cheng C. Heat flow and distribution during induction of general anesthesia. Anesthesiology. 1995 Mar;82(3):662-73. doi: 10.1097/00000542-199503000-00008. PMID 7879935
- [Background] Flynn MD, Sandeman DD, Mawson DM, Shore AC, Tooke JE. Cyclical hypothermia: successful treatment with ephedrine. J R Soc Med. 1991 Dec;84(12):752-3. doi: 10.1177/014107689108401224. No abstract available. PMID 1774760
- [Background] Sarti A, Recanati D, Furlan S. Thermal regulation and intraoperative hypothermia. Minerva Anestesiol. 2005 Jun;71(6):379-83. PMID 15886605
- [Background] Im UJ, Lee DJ, Kim MC, Lee JS, Lee SJ. Difference in Core temperature in response to propofol-remifentanil anesthesia and sevoflurane-remifentanil anesthesia. Korean J Anesthesiol. 2009 Dec;57(6):704-708. doi: 10.4097/kjae.2009.57.6.704. PMID 30625952
- [Background] Nakasuji M, Nakamura M, Imanaka N, Tanaka M, Nomura M, Suh SH. Intraoperative high-dose remifentanil increases post-anaesthetic shivering. Br J Anaesth. 2010 Aug;105(2):162-7. doi: 10.1093/bja/aeq121. Epub 2010 Jun 10. PMID 20542888
- [Result] Jo YY, Kim JY, Kim JS, Kwon Y, Shin CS. The effect of ephedrine on intraoperative hypothermia. Korean J Anesthesiol. 2011 Apr;60(4):250-4. doi: 10.4097/kjae.2011.60.4.250. Epub 2011 Apr 26. PMID 21602974